CLINICAL TRIAL: NCT04938388
Title: Comparison of Oral Semaglutide With Matched Oral Semaglutide Placebo as an Early Treatment for Latino Adults With Type 2 Diabetes Receiving Enhanced Lifestyle Care
Brief Title: Comparison of Oral Semaglutide w/ Placebo- Treatment for Latino Adults w/T2 Diabetes Receiving Enhanced Lifestyle Care
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator no longer at study site.
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Kristin Castorino, DO, Senior Research Physician, Sansum Diabetes Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: U1111-1238-3149
Record Dates: First submitted 2021-06-15; First posted 2021-06-24 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2; Glucose Metabolism Disorders (Including Diabetes Mellitus)
Keywords: Minority Health; Plants, Edible
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Single center, 56-week, randomized controlled, parallel group, double blind study comparing OS (active group) with Placebo (control group) in adult Latinos with established type 2 diabetes treated with usual diet/exercise modification alone and/or Metformin at randomization, with both groups under the supervision of the licensed SDRI study physician/Co-Investigator and also receiving enhanced lifestyle care.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Semaglutide (OS) with Enhanced Lifestyle Care (organic vegetables) (Active Comparator): Participants will start at a 3 mg dose of OS. If this minimum dose is not tolerated, the participant will be withdrawn from the study. After 4 weeks, the OS dose will be adjusted to 7 mg. After a further 4 weeks of study and thereafter, the OS dose will be adjusted at the study physician's discretion to 14 mg. At each study visit, the current dose of OS will be maintained, unless participants report moderate-to-severe nausea or vomiting for 3 or more days in the week before the scheduled visit. If participants report moderate-to-severe nausea or vomiting, the OS dose will be maintained or decreased at the study physician's discretion.
  Participants will be instructed to swallow the OS tablet whole (not crushed, cut or chewed) in the morning, in a fasted state, with up to 120 mL of plain water, at least 30 minutes before any other food, beverage, or oral medication.
  Interventions: Drug: Semaglutide Pill; Dietary Supplement: Fresh organic vegetables
- Oral Semaglutide (OS) Placebo with Enhanced Lifestyle Care (organic vegetables) (Placebo Comparator): Participants will start at a 3 mg dose of OS matched Placebo. If this minimum dose is not tolerated, the participant will be withdrawn from the study. After 4 weeks, the Placebo will be adjusted to 7 mg. After a further 4 weeks of study and thereafter, the Placebo will be adjusted at the study physician's discretion to 14 mg. At each study visit, the current dose of Placebo will be maintained, unless participants report moderate-to-severe nausea or vomiting for 3 or more days in the week before the scheduled visit. If participants report moderate-to-severe nausea or vomiting, the Placebo will be maintained or decreased at the study physician's discretion.
  Participants will be instructed to swallow the matched OS Placebo whole (not crushed, cut or chewed) in the morning, in a fasted state, with up to 120 mL of plain water, at least 30 minutes before any other food, beverage, or oral medication.
  Interventions: Dietary Supplement: Fresh organic vegetables

INTERVENTIONS:
Drug: Semaglutide Pill — All participants will start at a 3 mg dose of OS or matched Placebo. If this minimum dose is not tolerated, the participant will be withdrawn from the study. After 4 weeks, the OS dose (or Placebo) will be adjusted to 7 mg. After a further 4 weeks of study and thereafter, the OS dose (or Placebo) will be adjusted at the study physician's discretion to 14 mg. At each study visit, the current dose of OS (or Placebo) will be maintained, unless participants report moderate-to-severe nausea or vomiting for 3 or more days in the week before the scheduled visit.
  Other Names: Semaglutide 3 mg; Semaglutide 7 mg; Semaglutide 14 mg
  Arms: Oral Semaglutide (OS) with Enhanced Lifestyle Care (organic vegetables)
Dietary Supplement: Fresh organic vegetables — Prescriptions of organic vegetables

SUMMARY:
Researchers at Sansum Diabetes Research Institute want to learn more about how taking a new approved drug called oral Semaglutide, while eating fresh vegetables, impacts health in Hispanic/Latino adults with type 2 diabetes. This study drug is approved by the United States Food and Drug Administration and may be available by prescription for type 2 diabetes. To do this, 100 Hispanic/Latino adults who have type 2 diabetes will be split into two groups. Over one year, one group will take Semaglutide pills and the other group will take a placebo (a dummy pill that looks just like the real Semaglutide pill but does not contain the active drug). Neither the participants nor the study investigator nor the study doctor will know who is taking the real pill and who is taking the placebo. In case of an emergency, however, the study investigator and doctor can get this information. All participants will receive pills and vegetables every two weeks, have their health assessed by study staff, and meet with the study doctor six times over the course of the study. Participant weight, height, waist circumference, blood pressure, and blood glucose levels will be measured. Participants will also wear monitors to measure blood glucose, physical activity and sleep. Study staff will also ask questions about participant health, medications, mood, sleep, pain, exercise, diet, acculturation, household, language, and trust in doctors.

DETAILED DESCRIPTION:
Oral Semaglutide is the first oral formulation of a glucagon-like peptide-1 (GLP-1) receptor agonist developed for the treatment of type 2 diabetes (T2D). Monotherapy with once-daily oral Semaglutide has been shown to provide superior and dose-dependent decreases in HbA1c compared with placebo, and superior decreases in bodyweight in patients with T2D whose glycaemia was insufficiently controlled on diet and exercise. Recently, in patients with T2D and chronic kidney disease, Semaglutide was also effective in improving glycemic control and bodyweight with a low risk of hypoglycemia compared to placebo. Oral Semaglutide has also been shown to be superior to Sitagliptin. Results from the PIONEER 6 trial showed that no increased risk for major cardiovascular events was observed with oral Semaglutide in patients with T2D at high cardiovascular (CV) risk. In that study, Semaglutide reduced CV death and all- cause mortality by nearly 50% versus placebo after a median follow-up of 15.9 months. Therefore based on the evidence from the PIONEER trials, oral Semaglutide is likely to offer significant benefits for adults with T2D.

However in the United States (US), members of racial and ethnic minority groups are disproportionally affected by T2D and there is a paucity of information on what the potential impact of novel therapies such as oral Semaglutide might be for these populations. For example, the prevalence of both diagnosed and undiagnosed T2D is nearly twice as high among Mexican- origin Hispanic/Latino (hereafter Latino) adults compared to non-Latino whites. Likewise, rates of diabetes-related complications (including premature death from diabetes, acute stroke and end- stage renal disease) are also higher among Latino adults compared to their non-Latino white counterparts. For Latinos and other US minorities, beyond genetics and biological factors, it is recognized that sociocultural influences are also important factors in determining an individual's response to a therapy. In addition, self-identified race correlates with ancestry, which determines genomic variation, but this does not necessarily predict the response to a particular drug, nor can it be assumed that responses are similar between different races. As a corollary, being uninsured or a Medicaid recipient presents formidable challenges to improving cost-effective outcomes for people with diabetes. Currently, in the US, more than 29 million people are uninsured, with substantial inequalities in access to health care along economic, gender, racial, and ethnic lines. Racial and ethnic minority groups in the US also receive lower quality of health care compared with their white counterparts and disparities exist in the burden and cost of diabetes care for Medicare recipients. Identifying sub-groups with especially high risk of complications early in the course of T2D will also help clinicians to offer more cost-effective therapies. In addition, regulatory and policy decisions are increasingly based on a continuum of data from intensively monitored randomized clinical trials (RCTs) to real-world evidence (RWE), i.e., from tightly controlled, homogeneous populations to broader ones seen in usual clinical practice.

US minorities commonly live in "poorer" neighborhood environments with respect to access to healthy food sources, places to exercise or safety from crime. Plant-based dietary foods have the potential to help manage several major chronic diseases, including T2D. For underserved populations with T2D, food insecurity and low socioeconomic status are frequent barriers to nutrition-based self-management.

As a consequence, Sansum Diabetes Research Institute (SDRI) has recently created Farming for Life, which provides medically prescribed produce to Latino adults with non-insulin treated T2D. Farming for Life uses prescriptions of predominantly organic vegetable produce, as studies have shown that organic crops have higher concentrations of antioxidants and a lower incidence of pesticide residues than non-organic crops. There is growing evidence of an association between pesticide exposure and T2D risk.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ≥ 18 years of age at enrollment.
2. Self-reported Hispanic/Latino heritage.
3. Established diagnosis of T2D for at least 3 months prior to enrollment date.
4. HbA1c > 7.5% and ≤ 10.0% (58-86 mmol/mol) within the previous 6 months.
5. T2D treated with lifestyle alone or lifestyle + Metformin within the past 6 months prior to screening.
6. Ability to provide informed consent before any trial-related activities. Trial-related activities are any procedure that would not have been performed during normal management of the subject.
7. Based on the research staff's judgment, participant or participant's representative must have a good understanding, ability, and willingness to adhere to the protocol, including performance of self-monitored data collection during the wearable device portion of the study.

Exclusion Criteria:

1. Type 1 diabetes or a history of diabetic ketoacidosis.
2. T2D treated with oral medicines other than Metformin or any injectable GLP-1 receptor agonist or insulin within the past 6 months prior to screening.
3. Life expectancy < 12 months.
4. Any active clinically significant physical or mental disease or disorder which, in the investigator's opinion, could interfere with the participation in the study.
5. History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g., subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
6. Untreated pre-proliferative or proliferative retinopathy or maculopathy due to diabetes.
7. Renal impairment, defined as estimated glomerular filtration rate <30 mL/min/1.73 m2.
8. Personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia syndrome type 2.
9. Language barriers precluding comprehension of study activities and informed consent.
10. Participation in other research studies involving medication or device within 1 month prior to enrollment.
11. Known or suspected abuse of alcohol, narcotics, or illicit drugs.
12. Known or suspected allergy to OS, excipients, or related products.
13. Previous participation in this trial whether screened or randomized.
14. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures.
15. The receipt of any investigational drug (within 12 months) prior to this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-29 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
HbA1c < 7.0% | At 50 weeks
  proportion of participants achieving an HbA1c < 7.0% at 50 weeks post-baseline in both groups (OS versus Placebo) with both groups receiving enhanced lifestyle care.

SECONDARY OUTCOMES:
HbA1c | At 50 weeks
  Comparison with baseline (-2 weeks)
Weight | At 50 weeks
  Comparison with baseline (-2 weeks)
Waist circumference | At 50 weeks
  Comparison with baseline (-2 weeks)
Lying and standing blood pressure | At 50 weeks
  Comparison with baseline (-2 weeks)
Fasting glucose levels | At 50 weeks
  Comparison with baseline (-2 weeks)
Fasting insulin levels | At 50 weeks
  Comparison with baseline (-2 weeks)
Calculation of insulin resistance (HOMA-B and HOMA-IR) | At 50 weeks
  Comparison with baseline (-2 weeks)
Lipid Levels | Comparison with baseline (-2 weeks) and at 50 weeks
  Lipid levels- (total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides)
Liver Function Test | Comparison with baseline (-2 weeks) and at 50 weeks
  Liver Function Test (AST, ALT, Albumin)
CGM Time In Range | Weeks 48-49
  Comparison of Continuous Glucose Monitoring data collected over weeks 48-49 with baseline of time in range (70-180 mg/dl) using continuous glucose monitoring
Number of Pill Counts | Comparison at 4, 8, 22, 34, and 48 weeks
  Adherence to prescribed medicines- Number of Pill Counts
Additional glucose-lowering medication (rescue medication) | Comparison at 4, 8, 22, 34, and 48 weeks
  The need for additional glucose-lowering medication (rescue medication) initiated by the study physician with recording of additional medication by medication name
Number of participants with treatment-related adverse events assessed by research physician classified according to Good Clinical Practice guidelines | Data captured at baseline
  Participants unable to tolerate the treatment medication

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States